CLINICAL TRIAL: NCT05092542
Title: Multilevel Community-Based Mental Health Intervention to Address Structural Inequities and Adverse Disparate Consequences of COVID-19 Pandemic on Latinx Immigrant and African Refugees
Brief Title: Intervention to Address Disparate Mental Health Consequences of COVID-19 Pandemic on Latinx and African Newcomers
Acronym: RIWP+
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 07521; R01MH127733 (NIH)
Record Dates: First submitted 2021-10-22; First posted 2021-10-25 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Mental Health Issue; Mental Health Disorder; Stress, Emotional; Economic Problems
Keywords: Latinx immigrant; African refugee
MeSH Terms: conditions — Mental Disorders; Stress, Psychological

STUDY DESIGN:
Intervention Model Description: By including 240 Latinx immigrants and 60 African refugees recruited from CBO partners who are randomly assigned to treatment-as-usual CBO involvement or the RIWP intervention and a random sample comparison group of 900 Latinx immigrants, this mixed methods longitudinal waitlist control group design study with five time points over 28 months will test the effectiveness of the RIWP intervention and engagement with CBOs to reduce psychological distress, daily stressors, and economic precarity and increase protective factors (social support, critical awareness of/access to resources, English proficiency, cultural connectedness, and mental health service use).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Random Sample of Latinx Immigrants (No Intervention): random sample comparison group of Latinx immigrants who are NOT randomly assigned to a treatment condition
- Refugee & Immigrant Well-being Project (RIWP) Intervention (Experimental): 6-month mental health intervention that pairs university students with newcomers to engage in mutual learning, resource mobilization, and social change efforts
  Interventions: Behavioral: Refugee and Immigrant Well-being Project (RIWP)
- Treatment-as-usual Waitlist Control Group (No Intervention): participants recruited from community-based organizations receive usual services from community-based organizations and may participate in RIWP intervention in Year 3

INTERVENTIONS:
Behavioral: Refugee and Immigrant Well-being Project (RIWP) — 6-month mental health intervention that pairs university students with newcomers to engage in mutual learning, resource mobilization, and social change efforts
  Other Names: Refugee Well-being Project (RWP); Immigrant Well-being Project (IWP)
  Arms: Refugee & Immigrant Well-being Project (RIWP) Intervention

SUMMARY:
This study tests the effectiveness of a community-based peer advocacy, mutual learning, and social support intervention (Refugee and Immigrant Well-being Project) to reduce several negative consequences of the COVID-19 pandemic that are disproportionately impacting Latinx and Black populations: psychological distress, financial problems, and daily stressors. In partnership with five community-based organizations that focus on mental health, legal, education, and youth issues with Latinx immigrants and African refugees, we will also be able to examine the effects of people's involvement with community-based organizations and local and state policy changes on their mental health, economic stability, stressors, and social support. This is important not only for Latinx and Black populations and the large number of immigrants and refugees in the United States and worldwide, but also because the intervention model and what we learn from this study have the potential to alleviate mental health disparities experienced by other marginalized populations who face unequal access to social and material resources, disproportionate exposure to trauma and stress, and worse consequences of the COVID-19 pandemic.

DETAILED DESCRIPTION:
The goal of this study is to test a multilevel approach to reduce adverse consequences of the COVID-19 pandemic with disparate impacts on Latinx and Black immigrants and refugees by observing and implementing three nested levels of intervention: 1) an efficacious 6-month peer advocacy and mutual learning model (Refugee and Immigrant Well-being Project, RIWP); 2) engagement with community-based organizations (CBOs); and 3) structural policy changes expected to be enacted in response to the pandemic, such as a state disaster relief proposal for mixed status Latinx families and expanded statewide health insurance coverage. This community-based participatory research (CBPR) study builds on a long-standing collaboration with five community-based organizations (CBOs) that focus on mental health, education, legal issues, and system change efforts to improve the well-being of Latinx immigrants and African refugees. By including 240 Latinx immigrants and 60 African refugees recruited from CBO partners who are randomly assigned to treatment-as-usual CBO involvement or the RIWP intervention and a random sample comparison group of 900 Latinx immigrants, this mixed methods longitudinal waitlist control group design study with five time points over 28 months will test the effectiveness of the RIWP intervention and engagement with CBOs to reduce psychological distress, daily stressors, and economic precarity and increase protective factors (social support, critical awareness of/access to resources, English proficiency, cultural connectedness, and mental health service use). This study will also test the ability of the RIWP intervention and engagement with CBOs to increase access to the direct benefits of structural interventions (local/state relief-related policies) for Latinx and Black immigrants and refugees. Mechanisms of intervention effectiveness will be explored by testing mediating relationships between primary outcomes and protective factors. Investigators will also track local/state policy changes and obtain preliminary quantitative estimates of effects of these structural interventions on psychological distress, stressors, and economic precarity using propensity score matching. Qualitative interview data from a purposive subsample of participants and CBO staff will enable additional exploration of mechanisms of change, the effects of policy interventions on individuals, how CBOs contribute to enacting policies and helping people benefit from them, and the context of RIWP implementation at each site. This research is innovative and significant because it employs cutting-edge research design and intervention strategies to advance the science of multilevel mental health interventions that aim to understand and address underlying structural inequities and resulting mental health disparities that have been highlighted and exacerbated by the pandemic. Thus, this study will contribute not only to reducing the disparate adverse mental health, behavioral, and socioeconomic consequences of the COVID-19 pandemic but also to eliminating mental health disparities among Latinx and Black populations.

ELIGIBILITY:
Inclusion Criteria:

* All Latinx immigrants and African refugees aged 18 and older residing in New Mexico will be eligible to participate.

Exclusion Criteria:

* For the random sample of 1000 Latinx immigrants, exclusion criteria will be having used the services of one of the four community-based partner organizations serving Latinx immigrants within the past year (at time of study enrollment). For the 240 Latinx immigrants and 60 African refugees recruited through the five community-based organizations, exclusion criteria will be severe cognitive functioning problems or mental illness that is so severe as to impede participation in a group and that warrants immediate individual treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1212 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Psychological Distress | All 7 timepoints over 36 months
  DSM Level 1 Cross-Cutting Symptom Measure-Adult and COVID-19 and Mental Health Impacts Scale (from PhenX Toolkit)
Psychological Distress | All 7 timepoints over 36 months
  PHQ-9
Psychological Distress | All 7 timepoints over 36 months
  GAD-7
Physical Health | All 7 timepoints over 36 months
  WHODAS-2
Daily Stressors | All 7 timepoints over 36 months
  Perceived Stress Scale
Economic Precarity | All 7 timepoints over 36 months
  Job Insecurity General Social Survey 2018 Questions and RAND American Life Panel Impacts of COVID-19 Survey

SECONDARY OUTCOMES:
Access to Resources | All 7 timepoints over 36 months
  Satisfaction with Resources Scale
Social Support | All 7 timepoints over 36 months
  Medical Outcomes Study Social Support Survey, 8-item version
Cultural Connectedness | All 7 timepoints over 36 months
  Language, Identity, and Behavior Acculturation Scale
Health Services Use | All 7 timepoints over 36 months
  Composite International Diagnostic Interview (selected questions)
English Proficiency | All 7 timepoints over 36 months
  4 items about understanding, reading, speaking, and writing
Discrimination | All 7 timepoints over 36 months
  Experience of Discrimination (EOD) Scale

CONTACTS AND LOCATIONS:
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: Yes
After all analyses are completed and presentations/publications are finalized, a de-identified dataset will be available to other researchers, communities, or providers, upon request. All requests would have to be approved by the Community Advisory Council and would have to demonstrate that the proposed use of the data would contribute to the reduction of mental health disparities (e.g., through improved detection, diagnosis, treatment or prevention of mental illness or through contributing to knowledge of these issues) and would not harm any individuals or communities (e.g., through naïve use of the data that might result in misrepresentation of the experiences of Latinx immigrants or African refugee individuals, families, or communities).
  Also, the data will be entered and available through the NIMH Data Archive.
Supporting Information: Study Protocol
Time Frame: Within 6 months of the end of data collection in Year 4
Access Criteria: The NDA provides basic descriptive and aggregate summary information for general public use. Such summary information may include summary counts and general statistics on completed assessment instruments. Access to subject level datasets submitted and stored in the NDA will only be provided for research purposes through the completion of the NDA Data Use Certification: OMB Control Number: 0925-0667. For the majority of the data available in the NDA, Data Use Certifications will only be accepted from researchers who are sponsored by an institution registered in the NIH's eRA Commons with an active Federal-wide Assurance issued through the Office for Human Research Protections (OHRP). Additionally, the application must include a reason for access related to scientific investigation, scholarship or teaching, or other form of research.
URL: https://s3.amazonaws.com/nda.nih.gov/Documents/NIMH+Data+Archive+Policy.pdf